CLINICAL TRIAL: NCT02918955
Title: Definitive Chemo-Radiotherapy With or Without Up-front Neck Dissection for Regionally Advanced Head and Neck Squamous Cell Carcinoma: A Phase III Multi-center Prospective Randomized Controlled Trial With Two Additional Observational Cohorts
Brief Title: Definitive Chemo-Radiotherapy for Regionally Advanced Head and Neck Cancer With or Without Up-front Neck Dissection
Acronym: UPFRONT-NECK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE 00733/16
Record Dates: First submitted 2016-09-21; First posted 2016-09-29 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Neoplasms
Keywords: head and neck cancer; radiotherapy; chemotherapy; neck dissection; surgery; quality of life; toxicity; oropharyngeal cancer; laryngeal cancer; hypopharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Radiotherapy; Drug Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm rA (randomized) (Active Comparator): Concomitant chemo-radiotherapy with early salvage neck dissection if less than complete clinical response
  Interventions: Radiation: radiotherapy; Drug: Chemotherapy (Cisplatin); Procedure: Early Salvage Neck Dissection in case of less than cCR (Arm A only)
- Arm rB (randomized) (Experimental): Up-front neck dissection followed by radiotherapy with concomitant chemotherapy based on the cT pN cM staging after surgery
  Interventions: Procedure: up-front neck dissection; Radiation: radiotherapy; Drug: Chemotherapy (Cisplatin)
- Arm oA (non-randomized) (Active Comparator): Concomitant chemo-radiotherapy with early salvage neck dissection if less than complete clinical response
  Interventions: Radiation: radiotherapy; Drug: Chemotherapy (Cisplatin); Procedure: Early Salvage Neck Dissection in case of less than cCR (Arm A only)
- Arm oB (non-randomized) (Experimental): Up-front neck dissection followed by radiotherapy with concomitant chemotherapy based on the cT pN cM staging after surgery
  Interventions: Procedure: up-front neck dissection; Radiation: radiotherapy; Drug: Chemotherapy (Cisplatin)

INTERVENTIONS:
Procedure: up-front neck dissection
  Arms: Arm oB (non-randomized); Arm rB (randomized)
Radiation: radiotherapy — 70 Gy in 35 fractions to the macroscopic disease 50 Gy in 25 fractions (if sequential boost) or 56 Gy in 35 fractions (if simultaneous integrated boost) to the elective volumes 66 Gy in 35 fractions to the post-operative region with lymphatic extracapsular extension (Arm B only)
Drug: Chemotherapy (Cisplatin) — 100 mg/m2 every three weeks during radiotherapy
  In Arm B, chemotherapy can be omitted in case of a cT1-2 primary and a surgical downstaged pN0-1 neck without lymphatic extracapsular extension.
Procedure: Early Salvage Neck Dissection in case of less than cCR (Arm A only) — Early salvage neck dissection in case of residual lymph node disease will be performed based on the response evaluation by MRI and PET/CT performed 3 and 4 months after the end of (chemo)radiotherapy, respectively (and additional diagnostic modalities if clinically indicated by the physician) and not more than 3 weeks after this post-radiotherapy evaluation.
  In Arm A, a successful early salvage neck dissection without the operation of the primary tumor in case of less than clinical complete response (cCR) will be considered a component of the multimodality treatment and not as a failure.
  Arms: Arm oA (non-randomized); Arm rA (randomized)

SUMMARY:
Treatment of regionally-advanced head and neck squamous cell carcinoma (HNSCC) requires a multidisciplinary approach with a combination of surgery, radiotherapy (RT) and chemotherapy. Due to these aggressive combined modalities, patients undergoing treatment and many survivors develop toxicities which impact quality of life (QoL) and sometimes lead to mortality.

Lymph node metastases of HNSCC are frequent and considered one of the most important prognostic factors, resulting in decreased survival by 50%. More than three decades, the optimal management strategy of node positive HNSCC was a key subject of debate. In summary, the current literature provides us two important findings: First, with the contemporary imaging and treatment modalities, there is no role of a planned neck dissection (ND) added to (chemo)radiotherapy ((C)RT) in terms of oncological outcome and survival. Second, with modern RT techniques, a tailored treatment followed after an up-front neck dissection (UFND) allows a significant reduction of treatment volumes and de-escalation of the dose to the neck, leading to reduction of treatment related toxicities.

In this study strategies with and without up-front neck dissection prior to chemo-radiotherapy will be compared.

DETAILED DESCRIPTION:
The main objective of this project is to test the hypothesis that the addition of UFND prior to (C)RT results in a significant reduction of treatment toxicities and improvement of QoL in regionally advanced (cN2-3) HNSCC through dose de-escalation and volume reduction of RT.

The primary endpoint of this trial is to evaluate the toxicity from the beginning of radiotherapy until 90 days after the end of the treatment. The incidence of acute and subacute toxicities higher than grade ≥3 (CTCAE v.4, except for Xerostomia, for which RTOG/EORTC scale will be used) will be compared between study arms. Secondary endpoints include the survival endpoints for both treatment modalities; i.e. loco-regional control, progression-free and overall survival. Assessment of QoL (EORTC QLQ-C30 + H&N43), late toxicity, surgical complications, cost-effectiveness and the need of feeding-tube will be a part of the final analysis of this trial.

Trial design: randomized multi-center open-label comparative one-staged phase III trial with a superiority design and the primary endpoint of highest grade radiation toxicity during and until 90 days after the completion of the treatment. Interventions in both arms of the trial are considered as standard treatments. No experimental diagnostic tools will be used during the trial. In addition to the randomized arms, two identical observational arms will be opened for the patients who are diagnosed before the activation of the randomized arms, and subsequently for those who refuse to be randomized. Their aim is to prospectively acquire high quality data for patients who refuse randomization. The observational and randomized cohorts will be analyzed separately for the pre-defined endpoints.

For the calculation of the sample size, grade ≥3 acute radiation toxicity in the CRT alone (Arm A) was assumed as 70% based on literature. For the primary endpoint, a follow-up period of 90 days after the last day of (C)RT is needed after the accrual of the last patient. However, 2 years of follow-up after (C)RT is needed for the secondary endpoints (exception: oncological outcome and survival will be calculated from the day of randomization in order to avoid immortal time bias). On this basis, sample size was calculated based on the Pearson chi-squared test and performed in Stata. Assuming a toxicity fraction of 70% for any grade 3 or higher toxicity in Arm A, a relative risk of 0.5 (35% in Arm B), a two-sided alpha of 0.05, a power of 80%, a drop-out rate of 5%, and an allocation ratio of 1 we calculated an overall sample size of 65. Expected accrual time is 3 years.

ELIGIBILITY:
1. Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.
2. Patient should not be a participant in any interventional clinical trial.
3. Age ≥ 18 years.
4. WHO/ECOG performance status 0-2 within 28 days prior registration.
5. Histopathologically confirmed, previously untreated HNSCC of the oropharynx, hypopharynx or larynx within 6 weeks (42 days) of registration.
6. No cT4 primary tumor destructing and/or breaching through bone and/or cartilage (cortical invasion only is still eligible).
7. Clinical Nodal stage (cN) of at least cN1.
8. No evidence of distant metastases (cM0). No synchronous second primary HNSCC at the time of diagnosis.
9. No synchronous or previous malignancies. Exceptions are adequately treated basal cell carcinoma or SCC of the skin, or in situ carcinoma of the cervix uteri or breast with a cancer-free follow-up time of at least 3 years, or other previous malignancy with a disease-free interval of at least 5 years.
10. No prior radiotherapy to the head and neck region (or any RT fields/volumes which may overlap with the intended therapy volumes).
11. No prior neck dissection or single lymph node excision is allowed.
12. History and physical examination by treating physician (head and neck surgeon, medical oncologist or radiation oncologist) within 28 days prior registration.
13. Patients must have clinically and/or radiological documented measurable disease. At least one site of disease must be unidimensionally measurable as per RECIST 1.1. All imaging studies for staging must be performed within 28 days prior to registration.
14. Imaging of the head and neck (CT with contrast, PET/CT and/or MRI) within 28 days prior to registration: A CT scan (as part of the PET/CT is also accepted), with contrast is mandatory unless contraindicated (e.g. contrast allergy, renal insufficiency etc.). Note that a PET/CT scan alone, unless performed with radio-opaque contrast material is not sufficient for the CT-based evaluation of the head and neck area.
15. PET/CT of the whole body within 28 days prior registration
16. QoL and toxicity evaluation completed within 28 days or at the time of registration. Exceptions: 1) Language problems or any health problems interfering with the QoL assessment. 2) Patients who want to be enrolled into the observational arms and refuse to take part in the QoL assessments.
17. Patients with a contraindication against neck dissection are not eligible (e.g. medical co-morbidities, positive lymph node conglomerates enclosing and infiltrating carotid artery or merging with the primary tumor)
18. The patient must be expected to withstand neck dissection and radiotherapy combined with cisplatin.
19. Preservation of the accessory nerve during neck dissection should be possible. Patients expected to have a permanent shoulder dysfunction because of a planned sacrifice of the accessory nerve are not eligible.
20. Laboratory requirements within 28 days prior to accrual:

    1. Adequate renal function: Serum creatinine ≤1.5 mg/dL and/or creatinine clearance >50 mL/min estimated within 28 days prior accrual
    2. Absolute neutrophil count (ANC) ≥1.0 x 109/L
    3. Platelet count ≥75 x 109/L
    4. Hemoglobin ≥10 g/dL or 6.2 mmol/L (Note: The use of transfusion to achieve Hgb ≥10 g/dL is acceptable)
    5. Bilirubin <1.5 times of upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 times of ULN.
21. Women are not breastfeeding. Women with Child-bearing potential and using effective contraception (see Section 5.6), and not pregnant and agree not to become pregnant during participation in the trial and 2 years after chemoradiotherapy. A negative pregnancy test before inclusion (within 28 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and 2 years after chemoradiotherapy.
22. No allergy to study drugs or to the excipients in their formulation.
23. No peripheral neuropathy ≥grade 2 according to CTCAE v4.03 (grade 2 = moderate symptoms limiting instrumental ADL)
24. No co-existing disease prejudicing survival (expected survival <6 months).
25. No severe cardiac illness: Myocardial infarction within 6 months prior to randomization, severe congestive heart failure, severe cardiomyopathy, ventricular arrhythmia, unstable angina, uncontrolled hypertension.
26. No active bacterial or fungal infection requiring intravenous antibiotics at the time of registration
27. No Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 28 days before registration.
28. No hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
29. No clinically manifested Acquired Immune Deficiency Syndrome (AIDS) or immune-compromised patients. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.

Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute & subacute toxicity based on CTCAE scoring system v4.03 | from the beginning of radiotherapy until 90 days after the end of the treatment

SECONDARY OUTCOMES:
Number of patients with late Toxicity based on CTCAE scoring system v4.03 | beginning from 91 days after the end of radiotherapy until the end of the 2 years follow up
Change from baseline quality of life(QoL)using EORTC QLQ-C30 v3&EORTC QLQ-H&N43 modules(Health related QoL specific for Head&Neck ca.)scores at end of RT, 3,12&24 months after RT.Swallowing (H&N43:4-item scale)3 months after RT is the primary QoL domain | up to 24-28 months depending on the treatment duration.
  EORTC QLQ-C30 and H&N43 will be used
Loco-regional control | 2 years from the randomization
Progression-free survival | 2 years from the randomization
Overall survival | 2 years from the randomization
Distant metastasis-free survival | 2 years from the randomization
Disease-specific survival | 2 years from the randomization
QoL comparison between the patients who accepted to be randomized (into rA and rB) and not (into oA and oB: in other words, patients who chose their own treatment strategy) | Baseline QoL and until the end of 2 years follow-up
Surgical complication rates | 2 years from the randomization
Rate of Isolated nodal control | 2 years from the randomization
  The absence of metastatic lymph node metastases in the neck without any synchronous or preceding local recurrence or distant metastases
Radiation dose and volumes | until the end of radiotherapy, expected to be on average 7 weeks
  The dose-volume histograms of all organs-at-risk (defined per protocol) will be compared between patients with and without up-front neck dissection. The doses will be reported in Gy and the volumes in cc.
Comparison of applied RT plan and the virtual RT plan done on the pre-UFND diagnostic CT images | until the end of radiotherapy, expected to be on average 7 weeks
  The dose-volume histograms of all organs-at-risk (defined per protocol) will be compared between the plans generated based on the pre- and post-UFND CT-scans of patients allocated the UFND arm. The doses will be reported in Gy and the volumes in cc.
Comparison between clinical and pathological stages of patients allocated to the UFND arm. according to the AJCC/UICC TNM staging system (7th edition). | until the generation of the definitive pathology report after the up-front neck dissection, expected to be within 3 weeks after patients' study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Olgun Elicin, MD, Study Chair — Department of Radiation Oncology, Inselspital
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern
  - University Hospital of Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No